CLINICAL TRIAL: NCT00909597
Title: A Multicenter, Randomized, Double Blind (Double Dummy), Active Controlled Study to Compare the Safety, Tolerability and Effect on Glycemic Control of Taspoglutide Versus Pioglitazone in Type 2 Diabetes Patients Inadequately Controlled on Therapy With Sulfonylurea or Metformin Plus Sulfonylurea
Brief Title: A Study of Taspoglutide Versus Pioglitazone in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BC21893; 2009-009157-24
Record Dates: First submitted 2009-05-27; First posted 2009-05-28 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pioglitazone; taspoglutide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- pioglitazone (Active Comparator)
  Interventions: Drug: pioglitazone
- taspoglutide 10mg (Experimental): taspoglutide 10mg sc weekly
  Interventions: Drug: taspoglutide
- taspoglutide 10mg/20mg (Experimental): taspoglutide 20mg sc weekly after 4 weeks of taspoglutide 10mg sc weekly
  Interventions: Drug: taspoglutide

INTERVENTIONS:
Drug: pioglitazone — 30mg po once daily for 4 weeks, followed by 45mg once daily
  Arms: pioglitazone
Drug: taspoglutide — 10mg sc once weekly
  Arms: taspoglutide 10mg
Drug: taspoglutide — 10mg sc once weekly for 4 weeks, followed by 20 mg sc once weekly
  Arms: taspoglutide 10mg/20mg

SUMMARY:
This double-blind, double-dummy 3 arm study will evaluate the efficacy, safety and tolerability of taspoglutide versus pioglitazone in patients with type 2 diabetes mellitus inadequately controlled with sulfonylurea monotherapy or sulfonylurea plus metformin combination therapy. After an initial screening period, patients will be randomized to one of 3 groups, to receive a)taspoglutide 10mg sc weekly, b)taspoglutide 20mg sc weekly after 4 weeks of taspoglutide 10mg sc weekly or c)pioglitazone 45mg/day po after 4 weeks of pioglitazone 30mg/day po.The anticipated time on study treatment is 24 months, and the target sample size is 500+ individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-75 years of age;
* type 2 diabetes mellitus;
* treated with stable sulfonylurea monotherapy or metformin + sulfonylurea for >=12 weeks prior to screening;
* HbA1c >=7.0% and <=10% at screening;
* stable weight +/-5% for >=12 weeks prior to screening.

Exclusion Criteria:

* type 1 diabetes, diabetes resulting from pancreatic injury, or secondary forms of diabetes;
* clinically significant diabetic complications;
* clinically symptomatic gastrointestinal disease;
* >3 episodes of severe hypoglycemia within 6 months before screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 756 (Actual)
Dates: Start 2009-05; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Absolute change from baseline in HbA1c | 24 weeks

SECONDARY OUTCOMES:
Proportion of patients achieving target HbA1c <=6.5%, <=7% | weeks 24, 52 and 104
Absolute/percentage change from baseline in body weight; responder rate for body weight; absolute/percentage change from baseline in waist and hip circumference;absolute/percentage change from baseline in fasting plasma glucose | weeks 24, 52 and 104
Adverse events; laboratory parameters; cardiovascular events | At each clinic visit up to 106 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (127):
- United States (55):
  - Buena Park, California
  - Chino, California
  - Los Angeles, California
  - Rancho Cucamonga, California
  - Roseville, California
  - Santa Ana, California
  - Chiefland, Florida
  - Coral Gables, Florida
  - Daytona Beach, Florida
  - Panama City, Florida
  - Port Charlotte, Florida
  - St. Petersburg, Florida
  - Winter Park, Florida
  - Atlanta, Georgia
  - Columbus, Georgia
  - Conyers, Georgia
  - Roswell, Georgia
  - Chicago, Illinois
  - Springfield, Illinois
  - Evansville, Indiana
  - Madisonville, Kentucky
  - Metairie, Louisiana
  - Bethesda, Maryland
  - Ayer, Massachusetts
  - Waltham, Massachusetts
  - Ferndale, Michigan
  - Minneapolis, Minnesota
  - Biloxi, Mississippi
  - Jackson, Mississippi
  - Olive Branch, Mississippi
  - Grand Island, Nebraska
  - Berlin, New Jersey
  - Brick, New Jersey
  - Toms River, New Jersey
  - Trenton, New Jersey
  - New York, New York
  - Staten Island, New York
  - Durham, North Carolina
  - Mooresville, North Carolina
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Bend, Oregon
  - Medford, Oregon
  - Beaver, Pennsylvania
  - Philadelphia, Pennsylvania
  - Scranton, Pennsylvania
  - Kingsport, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - Salt Lake City, Utah
  - South Burlington, Vermont
  - Richmond, Virginia
  - Spokane, Washington
  - Vancouver, Washington
  - Waukesha, Wisconsin
- Australia (2):
  - Camperdown, New South Wales
  - Wollongong, New South Wales
- Brazil (6):
  - Fortaleza, Ceará
  - Lago Sul, Federal District
  - Belo Horizonte, Minas Gerais
  - Marília, São Paulo
  - São Paulo, São Paulo
  - Sorocaba, São Paulo
- Canada (5):
  - Vancouver, British Columbia
  - Etobicoke, Ontario
  - London, Ontario
  - Thornhill, Ontario
  - Toronto, Ontario
- San José, Costa Rica
- France (7):
  - Besançon
  - Corbeil-Essonnes
  - Dommartin-lès-Toul
  - La Rochelle
  - Lille
  - Poitiers
  - Vénissieux
- Germany (9):
  - Berlin
  - Essen
  - Falkensee
  - Mainz
  - Münster
  - Rodgau
  - Siegen
  - Sulzbach-Rosenberg
  - Wangen
- Mexico (6):
  - Aguascaliente
  - Celaya
  - Cuernavaca
  - Guadalajara
  - Mexico City
  - Monterrey
- Auckland, New Zealand
- San Isidro, Peru
- Poland (4):
  - Gdansk
  - Krakow
  - Lublin
  - Wroclaw
- Rio Piedras, Puerto Rico
- Russia (7):
  - Moscow
  - Penza
  - S.Petersburg
  - Saint Petersburg
  - Saratov
  - Voronezh
  - Yaroslavl
- Slovakia (3):
  - Bratislava
  - Dolný Kubín
  - Levice
- Cape Town, South Africa
- Spain (5):
  - Almería, Almeria
  - Barcelona, Barcelona
  - Pamplona, Navarre
  - Oviedo, Principality of Asturias
  - Barakaldo, Vizcaya
- Thailand (3):
  - Chiang Mai
  - Pathum Thani
  - Songkhla
- Ukraine (3):
  - Kiev
  - Odesa
  - Vinnitsa
- United Kingdom (7):
  - Atherstone
  - Birmingham
  - Chesterfield
  - Dumfries
  - Glasgow
  - Hinckley
  - Reading